CLINICAL TRIAL: NCT04861480
Title: Phase I Clinical Study of CAR-T Cells (C-4-29) in the Treatment of Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Dual-target CAR-T Cells (C-4-29) in the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB04
Record Dates: First submitted 2021-04-06; First posted 2021-04-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-4-29 cells (Experimental): Infusion of C-4-29 cells by dose-escalating
  Interventions: Biological: C-4-29 Cells

INTERVENTIONS:
Biological: C-4-29 Cells — Drug: C-4-29 Cells； Administration method: intravenous infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This is a phase I clinical study to evaluate the safety and tolerability of C-4-29 in patients with relapsed or refractory multiple myeloma, and to obtain the maximum tolerated dose of C-4-29 and phase II Recommended dose.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label study. The study plans to set up 3 dose groups, adopting a dose-escalating 3+3 design, and plan to recruit about 9-18 subjects with relapsed or refractory multiple myeloma.C-4-29 cells will be infused to the subject by intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, no gender limit;
2. Diagnosed with multiple myeloma according to the IMWG diagnostic criteria.
3. Received third-line and above regular treatments (including proteasome inhibitors or immunomodulators) that are ineffective or intolerable;
4. The disease is measurable during screening:

   1. Serum M protein level ≥0.5g/dL, or urine M protein level ≥200mg/24h;
   2. Or light chain type MM with undetectable serum or urine disease: serum immunoglobulin free light chain ≥10mg/dL and serum immunoglobulin κ/γ free light chain ratio is abnormal;
   3. Or evaluable extramedullary lesions with the largest transverse diameter ≥ 1 cm.
5. ECOG 0～2 points;
6. The expected survival time is more than 12 weeks;
7. No serious mental disorders;
8. The function of important organs is basically normal:

   1. Heart function: echocardiography indicates that the cardiac ejection fraction is ≥50%, and the electrocardiogram has no obvious abnormalities;
   2. Renal function: serum creatinine≤2.0×ULN;
   3. Liver function: ALT and AST ≤3×ULN;
   4. Total bilirubin and alkaline phosphatase≤2×ULN (Gilbert syndrome≤3.0×ULN);
   5. Blood oxygen saturation>92%.
9. Have standards for apheresis or venous blood collection, and no other cell collection contraindications;
10. The subject agrees to use reliable and effective contraceptive methods for contraception within 1 year after signing the informed consent form to receiving C-4-29 cell infusion (excluding safe period contraception).
11. The patient himself or his guardian agrees to participate in the clinical trial and signs the ICF, indicating that he understands the purpose and procedures of the clinical trial and is willing to participate in the research.

Exclusion Criteria:

1. Have received CAR-T therapy or other genetically modified cell therapy;
2. With central nervous system disease at the time of screening ;
3. Participated in other clinical studies within 1 month before screening;
4. Have received a live attenuated vaccine within 4 weeks before screening;
5. Have received the following anti-tumor treatments before apheresis: received chemotherapy, targeted therapy or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter);
6. Within 7 days before apheresis, there are active infections or uncontrollable infections that require systemic treatment (except CTCAE grade 1 genitourinary system infection and upper respiratory tract infection);
7. Suffered from plasma cell leukemia at the time of screening ;
8. Suffered from other malignant tumors other than multiple myeloma within 3 years before screening, except for the following cases: malignant tumors that have received radical treatment, and there is no known active disease for ≥3 years before enrollment; or fully treated non-melanoma skin cancer with no evidence of disease;
9. Except for hair loss or peripheral neuropathy, the toxicity of previous anti-tumor treatments has not improved to the baseline level or ≤grade 1;
10. Subjects who have received systemic steroid treatment within 7 days before apheresis or who have been determined by the investigator to require long-term systemic steroid treatment during treatment (except for inhaled or topical use);
11. Suffered from any of the following heart diseases:

    1. NYHA stage III or IV congestive heart failure;
    2. Myocardial infarction or CABG occurred ≤6 months before enrollment;
    3. Clinically significant ventricular arrhythmia, or history of unexplained syncope (except for cases caused by vasovagal or dehydration);
    4. History of severe non-ischemic cardiomyopathy.
12. Active autoimmune diseases;
13. HBsAg or HBcAb positive and HBV DNA is greater than the normal range; HCV antibody is positive and HCV RNA greater than the normal range; HIV antibody positive; syphilis positive; CMV DNA positive;
14. Have experienced a venous embolism event (for example: pulmonary embolism or deep vein thrombosis) and requires anticoagulation therapy or the subject meets the following conditions: a. Bleeding of grade 3 to 4 lasting more than 30 days; b. Have sequelae caused by venous thrombosis (such as persistent dyspnea and hypoxia);
15. Women who are pregnant or breastfeeding, and male or female subjects who plan to have children within 1 year after receiving C-4-29 cell reinfusion;
16. Other situations considered by the researcher to be unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after C-4-29 infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of C-4-29 cells[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Objective response rate after C-4-29 infusion [Effectiveness] | 3 months
  Objective response rate includes sCR, CR, VGPR, PR, MR
AUCS of C-4-29 cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 28 days
CMAX of C-4-29 cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of C-4-29 cells expanded in peripheral blood
TMAX of C-4-29 cells [Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Peripheral blood M protein contents after C-4-29 infusion [Cell dynamics] | 3 months
  Periodic detection of Peripheral blood M protein after cell infusion
Urine Bence-Jones protein contents after C-4-29 infusion [Cell dynamics] | 3 months
  Periodic detection of Urine Bence-Jones protein after cell infusion
Immunogenicity of C-4-29 cells | 3 months
  Anti-CAR antibody

OTHER OUTCOMES:
Overall survival after C-4-29 infusion | 2 years
  OS is defined as the time from C-4-29 cell infusion to death due to any cause
Progression-free survival after C-4-29 infusion | 2 years
  PFS is defined as the time from the start of the C-4-29 infusion to the first disease progression or death from any cause
Duration of relief after C-4-29 infusion | 2 years
  DOR is defined as the time from reaching MR or better to disease progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China